CLINICAL TRIAL: NCT00934778
Title: Evaluation of Two Minimally Invasive Endoscopic Techniques for the Diagnosis of the Diffuse Lung Diseases.
Brief Title: Minimally Invasive Endoscopy in Diffuse Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09/H0708/18
Record Dates: First submitted 2009-06-12; First posted 2009-07-08 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Lung Disease; Lung Cancer
Keywords: Confocal microscopy; Endocytoscopy; Diffuse lung disease; Minimally invasive; Lung cancer and dysplasia
MeSH Terms: conditions — Lung Diseases; Lung Neoplasms | interventions — Microscopy, Confocal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bronchoscopy (Experimental)
  Interventions: Procedure: Confocal microscopy and endocytoscopy

INTERVENTIONS:
Procedure: Confocal microscopy and endocytoscopy — 2 probe based imaging systems for use via the working channel of the bronchoscope. 0.5ml of methylene blue injected into airways for endocytoscopy. Each procedure takes about 2-3 minutes.

SUMMARY:
We want to compare 2 new systems for obtaining very detailed images of the smallest airways, in the hope that they can be used to provide useful information about lung diseases without the need for invasive tests.

Two new systems have been developed for use down the bronchoscope, which provide video imaging of the smallest airways, each system looking at a different aspect of the structure of the airway walls. In principal, this method could provide useful information which may reduce the need for a surgical lung biopsy. We will therefore be assessing the value of the additional information obtained with these two new systems.

The purpose of this research project is to gather information using both systems to gain a greater understanding of the tissue characteristics of various diseases without the need for a biopsy.

DETAILED DESCRIPTION:
Diffuse lung disease (DLD) remains a challenging area for diagnosis and treatment. Features suggestive of the various histological subtypes of DLD can be obtained from the clinical history and examination, and can also seen on cross-sectional imaging (high resolution computed tomography (HRCT) scanning), however final diagnosis very often relies on the results of more invasive testing. The gold-standard diagnostic tool is the surgical lung biopsy, but this requires a general anaesthetic and either thoracoscopy or thoracotomy. The morbidity and even mortality attached to this approach in these patients, many of whom have significant respiratory compromise, has resulted in less invasive techniques being employed in many instances. At present, this involves the use of bronchoalveolar lavage (BAL) and transbronchial biopsies via the fibreoptic bronchoscope. BAL can be distressing for patients if there is spill-over of lavage fluid into the larger airways, and transbronchial biopsies lead to significant bleeding or pneumothorax in around 5% of patients. Even with biopsies and BAL, some patients still progress to surgical lung biopsy.

There have recently been developed 2 systems for use via the working channel of the endoscope which provide imaging of the distal airways and alveoli in vivo and in real time. These are described below. In principal, these could provide diagnostic information in the setting of DLD without the need for biopsies or BAL, reducing morbidity and cost associated with sample processing, and shortening the time to diagnosis. The ideal situation would be that sufficient morphological and histological information could be obtained using these systems, thus obviating altogether the need for surgical biopsy in this patient group, providing further benefits for the patient and potentially huge cost savings for institutions.

Cellvizio® Lung (Mauna Technology) Confocal microscopy is the standard tool for ultrahigh resolution imaging in biomedical research. Mauna Technology has developed a 1.4mm diameter Alveoflex Confocal Miniprobe™ which can be deployed down the working channel of a standard bronchoscope. Elastin is the main in vivo fluorophore, and images are acquired by gentle contact, providing microstructural detail of the alveolus on multiple tissue layers. Because the system takes advantage of the natural fluorescence of the lung tissues, no patient preparation is required.

Endocytoscope system (ECS) The endocytoscope is a newly developed system that can be passed through the working channel of a standard bronchoscope, and provides high magnification views (x450) of cell surfaces. About 5mls of 0.5% methylene blue solution is used to stain the area of interest, and images are obtained by contact with the cell surface. Use of the ECS has already been shown to allow discrimination between normal and abnormal tissue in situ in the setting of bronchial dysplasia and malignancy.

Aim of research The purpose of this research project is to build up a database of information gathered using both systems so that features correlating with the different diffuse lung diseases (e.g. sarcoidosis, interstitial pneumonias, drug induced lung diseases, emphysema) can be recorded. Patients with normal lung parenchyma and focal disease such as lung cancer will also be evaluated in order to develop a better understanding of pulmonary morphology using these techniques. By using two potentially complimentary systems that look at different structural aspects of the target tissues, a greater understanding of in vivo tissue characteristics can be gained. It is hoped that diagnostic criteria can then be drawn up for individual diseases that can then be assessed prospectively in trials.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 or over
* Scheduled for bronchoscopy as part of clinical care
* No bleeding diathesis or therapeutic anticoagulation

Exclusion Criteria:

* Unable to provide informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
To determine characteristic features of different lung disease on confocal microscopy and endocytoscopy. | Interim analysis every 20 cases

SECONDARY OUTCOMES:
Rate of complications and side-effects over and above standard bronchoscopy. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pallav Shah, MBBS, MD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust